CLINICAL TRIAL: NCT06633731
Title: Clinical Case Study Evaluating the Efficacy and Tolerability of a Topical Facial Treatment on Healthy Females with Fitzpatrick Skin Types V and VI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Collaborators: Tone Dermatology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS-2023-01
Record Dates: First submitted 2024-10-03; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Skin Smoothness; Radiance; Overall Appearance
Keywords: anti-aging; Fitzpatrick Skin Types V and VI; Skin Rejuvenation
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topical Treatment (Experimental): Subjects received a topical facial treatment applied by a license esthetician in a series of 3 sessions at 1 month intervals. The treatment included a topical treatment, biocellulose mask, and serum. Additionally, subjects followed a 12 weeks skincare regimen including a gentle cleanser, bland moisturizer, and bland sunscreen.
  Interventions: Other: Biocellulose Mask; Other: Post Procedure Cream; Other: Gentle Cleanser; Other: Facial Moisturizer; Other: sunscreen

INTERVENTIONS:
Other: Biocellulose Mask — Immediately after treatment, a Biocellulose Mask was applied to the subjects global face for 8 to 10 minutes.
Other: Post Procedure Cream — Immediately after treatment and after Biocellulose Mask removal, the Post-Procedure Cream was applied to the subjects global face. Subjects were instructed to apply to the global face from days 1 - 3 post treatment.
  Other Names: CMT Post Procedure Cream, Revision Skincare
Other: Gentle Cleanser — Subjects were instructed to wash their face with the Gentle Foaming Cleanser twice daily for 12 weeks.
  Other Names: Gentle Foaming Cleanser, Revision Skincare
Other: Facial Moisturizer — Subjects were instructed to apply the facial moisturizer twice daily to the global face from day 3 after treatment until next study visit.
Other: sunscreen — Subjects were instructed to apply the bland sunscreen to the global face once daily in the morning, with re-application with extended sun exposure per FDA guidelines.
  Other Names: Cetaphil® Sheer Mineral Sunscreen SPF 30

SUMMARY:
This single-center, open-label, clinical case trial was conducted to evaluate the efficacy and tolerability of a topical facial treatment when applied by a license esthetician in clinic in a series of 3 sessions with 1 month intervals on healthy women with Fitzpatrick Skin Types V and VI and mild to moderate global facial radiance, skin smoothness, and overall appearance. The treatment will include an topical facial treatment, biocellulose mask, and post-procedure cream. Furthermore subjects followed a 12 week skincare regimen consisting of a gentle cleanser, bland moisturizer, and bland sunscreen. Eleven (11) healthy female subjects completed the clinical study.

DETAILED DESCRIPTION:
This single-center, open-label, clinical case trial was conducted to evaluate the efficacy and tolerability of a topical facial treatment when applied by a license esthetician in clinic in a series of 3 sessions with 1 month intervals on healthy women with Fitzpatrick Skin Types V and VI and mild to moderate global facial radiance, skin smoothness, and overall appearance. The treatment will include an topical facial treatment, biocellulose mask, and post-procedure cream. Furthermore subjects followed a 12 week skincare regimen consisting of a gentle cleanser, bland moisturizer, and bland sunscreen. The efficacy and tolerability of the topical facial treatment in improving mild to moderate global facial radiance, skin smoothness, and overall appearance was evaluated by Investigator clinical efficacy grading and tolerability grading by a board-certified dermatologist, subject tolerability grading, and clinical photography.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Fitzpatrick Skin Type V and VI
* Individuals with mild to moderate global facial radiance, skin smoothness, and overall appearance (Score 2 - 6 on a 10-point modified Griffiths scale).
* Individuals willing to undergo a washout period of 3 days.

Exclusion Criteria:

* Individuals who are nursing (breastfeeding), pregnant, or planning to become pregnant during the study.
* Individuals currently having or having a history of cold sores (Herpes Simplex) on the face.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Change in Investigator Clinical Efficacy Grading versus Baseline | 12 weeks
  The primary efficacy endpoint will be favorable analysis of the Investigator Clinical Efficacy Grading of radiance, skin smoothness, and overall appearance using a Modified Griffith's 10-point scale at week 4, week 8, and week 12 versus baseline (0:None, 9=Severe). A reduction in score indicates improvement.
Lack of Significant Change in Investigator Tolerability Parameters versus Baseline | 12 weeks
  The primary tolerability endpoint will be favorable analysis of Investigator Tolerability grading of erythema, edema and dryness completed by study investigator at baseline, weeks 4, 8 and 12. Local cutaneous tolerability will assessed using a four-point scale: 0 = None 1 = Mild 2 = Moderate 3 = Severe. A decrease in score indicates an improvement.
Lack of Significant Change in Subjective Tolerability versus Baseline | 12 weeks
  The secondary tolerability endpoint will be favorable analysis of Subject Tolerability grading of burning, itching, and stinging completed by subjects at baseline, weeks 4, 8 and 12. Local cutaneous tolerability will assessed using a four-point scale: 0 = None 1 = Mild 2 = Moderate 3 = Severe. A decrease in score indicates an improvement.

SECONDARY OUTCOMES:
Clinical Photography: VISIA-CR and Antera 3D | 12 weeks
  The secondary efficacy endpoint will be favorable analysis of clinical photography including VISIA® and Antera 3D® digital imaging at week 4, 8, and 12 versus baseline. A reduction in visual radiance, skin smoothness, and overall appearance on post-baseline timepoints compared to baseline is indicated an improvement
Change in Facial Parameters in a Self-Assessment Questionnaire versus Baseline and Percent Agreement | 12 weeks
  The secondary endpoint will be favorable analysis of Self-Assessment Questionnaires completed by subjects at baseline, week 4, week 8, and week 12. Subjects are asked to rate statements based on a scoring system ranging from 5 (completely agree) to 1 (completely disagree). A change in response values at weeks 4, 8, and 12 compared to baseline response values indicates an improvement. The best outcome is to Completely Agree with the statement / question being asked.

CONTACTS AND LOCATIONS:
Locations (1):
- Tone Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No